CLINICAL TRIAL: NCT01154400
Title: Grant Title: Eicosapentaenoic Acid and Protein Modulation to Induce Anabolism in COPD
Brief Title: Hydrolyzed Casein and Whey Protein Supplementation and the Addition of Leucine to Induce Protein Anabolism in Malnourished COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 109237
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: casein protein; whey protein; hydrolysates; leucine; protein metabolism; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Caseins; Whey; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Casein protein hydrolysates (Experimental): 15 g casein protein hydrolysates and 15 g maltodextrin
  Interventions: Dietary Supplement: Casein protein hydrolysates
- Whey protein hydrolysates (Experimental): 15 g whey protein hydrolysates and 15 g maltodextrin
  Interventions: Dietary Supplement: Whey protein hydrolysates
- Casein protein hydrolysates + LEU (Experimental): 15 g casein protein hydrolysates + 2.1 g LEU (40% of EAA content) + 15 g maltodextrin
  Interventions: Dietary Supplement: Casein protein hydrolysates + LEU
- Whey protein hydrolysates + LEU (Experimental): 15 g whey protein hydrolysates + 1.5 g LEU (40% of EAA content) + 15 g maltodextrin
  Interventions: Dietary Supplement: Whey protein hydrolysates + LEU

INTERVENTIONS:
Dietary Supplement: Casein protein hydrolysates — 15 g casein protein hydrolysates + 15 g maltodextrin
  Other Names: Casein
  Arms: Casein protein hydrolysates
Dietary Supplement: Whey protein hydrolysates — 15 g whey protein isolate + 15 g maltodextrin
  Other Names: Whey
  Arms: Whey protein hydrolysates
Dietary Supplement: Casein protein hydrolysates + LEU — 15 g casein protein hydrolysate + 2.1 g LEU (40% of EAA content) + 15 g maltodextrin
  Other Names: Casein + LEU
  Arms: Casein protein hydrolysates + LEU
Dietary Supplement: Whey protein hydrolysates + LEU — 15 g whey protein isolate + 1.5 g LEU (40% of EAA content) + 15 g maltodextrion
  Other Names: Whey + LEU
  Arms: Whey protein hydrolysates + LEU

SUMMARY:
The aim of this study is the first aim of a NIH project that consists of 3 aims. The first aim examines the acute effects of two high-quality milk proteins (casein vs. whey) on whole-body and muscle protein metabolism in COPD patients with severe loss of muscle mass and the effects of adding leucine. The principal endpoints will be the extent of stimulation of net whole body protein synthesis as this is the principal mechanism by which either amino acid or protein intake causes muscle anabolism. After determining the optimal nutritional formulation based on the first aim we will continue to work on the second and third aim where fish oil supplementation will be part of the nutritional intervention as well.

DETAILED DESCRIPTION:
Cachectic COPD patients are characterized by a decreased muscle protein synthesis and an elevated myofibrillar protein breakdown. A substantial number of these patients, characterized by an enhanced systemic inflammatory response, fails to respond to nutritional therapy, which is of clinical relevance as weight gain to nutritional therapy is a significant, independent predictor of mortality in COPD.

In the present study, the acute protein anabolic effect of two high-quality milk protein supplements in COPD will be examined by comparing a hydrolyzed casein and whey protein meal. We make use of hydrolyzed proteins to correct for absorption differences. Furthermore the effects of these milk proteins with or without enrichment of leucine will be investigated.

Variables of interest are: net whole body protein synthesis; whole body protein synthesis and breakdown rate; whole body myofibrillar protein breakdown rate; whole body collagen breakdown; kinetics of insulin; glucose; amino acid levels.

It is the investigators hypothesis that a nutritional supplement containing casein protein and high levels of leucine will target the metabolic alterations of these cachectic COPD patients and will specifically stimulate protein anabolism. The knowledge gained from this study will benefit our insight in terms of promotion of protein anabolism in COPD patients. The long-term goal is to reformulate nutritional composition in accord with the effects of COPD on protein metabolism in order to ameliorate or even prevent progressive muscle wasting in these subjects, and improve their quality of life and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe chronic airflow limitation, defined as measured forced expiratory volume in one second (FEV1) ≤ 70% of reference FEV1
* Shortness of breath on exertion
* Age 45 years and older
* Clinically stable condition and not suffering from respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever) at least 4 weeks prior to the study
* Cachexia based on the criteria: Body mass index ≤ 25 kg/m2 and/or FFM-Index: FFM/height2 ≤ 17 (males), 15 (females) kg/m2 and/or recent involuntary weight loss

Exclusion Criteria:

* Established diagnosis of malignancy
* Presence of fever within the last 3 days
* Established diagnosis of Diabetes Mellitus
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
* Allergy to cow's milk protein
* Any other condition according to the PI or study physicians would interfere with proper conduct of the study / safety of the patient
* Failure to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in net whole body protein balance | 6 hours
  Net whole body protein synthesis before and after protein feeding

SECONDARY OUTCOMES:
Change in whole body protein synthesis rate | 6 hours
  Whole body protein synthesis before and after protein feeding
Change in whole body protein breakdown rate | 6 hours
  Whole body protein breakdown rate before and after protein feeding
Change in whole body collagen breakdown | 6 hours
  Whole body collagen breakdown before and after protein feeding
Change in insulin concentration | 6 hours
  Plasma insulin during protein feeding
Change in glucose concentration | 6 hours
  Plasma glucose concentration during protein feeding
Change in plasma amino acid levels | 6 hours
  Plasma amino acid level during protein feeding
Change in whole body myofibrillar protein breakdown rate | 6 hours
  Whole body myofibrillar protein breakdown before and after protein feeding

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Jonker R, Deutz NE, Erbland ML, Anderson PJ, Engelen MP. Hydrolyzed casein and whey protein meals comparably stimulate net whole-body protein synthesis in COPD patients with nutritional depletion without an additional effect of leucine co-ingestion. Clin Nutr. 2014 Apr;33(2):211-20. doi: 10.1016/j.clnu.2013.06.014. Epub 2013 Jul 1. PMID 23886411